CLINICAL TRIAL: NCT05897255
Title: Effects of SEMG Biofeedback With Core Muscle Strengthening Exercises and Kinesiotaping on Diastasis Recti in Post-partum Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUI/CTR/2023/7
Record Dates: First submitted 2023-05-31; First posted 2023-06-09 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-05

CONDITIONS: Diastasis Recti Abdominis

STUDY DESIGN:
Intervention Model Description: Parallel Group Randomized Control Trial
Who Masked: Participant
Masking Description: Participants will be unaware of the type of the intervention they would be receiving.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Active Comparator): In Control group, conventional method to reduce diastasis recti will be provided.
  Commonly used exercises in the treatment of DRA including abdominal hollowing, curl-ups, sit-ups, pelvic bridging, SLR will be performed by the patients.
  The conventional exercise program will be given 3days/week for 6 weeks and will include 2 sets of 5 reps of each exercise.
  Interventions: Device: Surface EMG Biofeedback
- Experimental Group A (Experimental): In experimental group A, Kinesiotape along with core strengthening exercises will be provided.
  The core strengthening exercise program will be given 45 minutes of session 3days/week for 6 weeks. Each exercise will have 5-10 repetitions with a period of rest in between to avoid fatigue and muscle spasm.
  Interventions: Device: Surface EMG Biofeedback
- Experimental Group B (Experimental): In experimental group B, SEMG biofeedback assisted core strengthening exercises with kinesiotaping will be provided.
  Surface EMG activity will be recorded from the left and right abdominal muscles while the exercises will be performed in different positions.
  Interventions: Device: Surface EMG Biofeedback

INTERVENTIONS:
Device: Surface EMG Biofeedback — Surface EMG activity will be recorded from the left and right abdominal muscles while the exercises will be performed in different positions. Electrical signals in the muscle are measured and displayed on the screen and are amplified into sounds that the patient can hear. This feedback increases patient effort and participation and provides the data and documentation required to measure patient outcomes and quantify progress. Electrical activity from Rectus Abdominis muscle, External Oblique muscle and Transversus Abdominis muscle will be recorded with their specific exercises. SEMG Biofeedback protocol of a series of ten second contractions, each contraction preceded by a ten second rest period will be followed. Starting with shorter work/rest periods as needed to build-up to these intervals are acceptable; for example, starting with 3-second contractions and 6-second rest periods, and then gradually increasing the duration of each.

SUMMARY:
Diastasis Rectus Abdominis is quite common during and after pregnancy. Abdominal core strengthening exercises have been proven to be very effective in reducing Inter rectus distance, however, the role of Biofeedback EMG assisted exercises in Diastasis Rectus have been poorly understood.

DETAILED DESCRIPTION:
This study is a Randomized Control Trial in which posr-partum females with diastasis recti will be recruited into a control and two experimental groups. In control group, patients will receive standard conservative treatment, whereas, in first experimental group, participants will receive core strengthening exercises with kinesiotaping; and in second experimental group, core strengthening exercises with kinesiotaping will be assisted by SEMG biofeedback. Patients will be evaluated pre and post-treatment for Inter rectus distance, abdominal strength and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Post-partum women aged 18-40 years
* Post-partum females from 6 to 24 months
* Diastasis rectus abdominus distance more than 2cm at any of 3 levels
* Primiparous or multiparous
* Spontaneous vaginal delivery and LSCS

Exclusion Criteria:

* Having skin sensitivity to taping
* Open abdominal wounds
* Abdominal skin diseases
* Abdominal hernia
* Other abdominal or back surgical history
* Any heart or respiratory conditions
* Neurological diseases

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female
Enrollment: 24 (Estimated)
Dates: Start 2022-08-11 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Inter Rectus Distance between rectus abdominis muscles. | 6 weeks
  We will measure the inter rectus distance by mechanical dial vernier caliper. It normally ranges between1 to 2cm at rest. Measurement of more than 2cm will confirm presence of diastasis rectus abdominis. IRD will be measured by instructing the patient to lie in hook line position, arms down by the side, with one pillow placed beneath the head. The examiner will palpate the medial and lateral borders of the right and left rectus abdominis muscle bellies at the marked locations of 2 cm above, below and at umbilicus levels.

SECONDARY OUTCOMES:
Abdominal Strength and core stability will be assessed by Mc Gill torso muscular endurance test battery. | 6 weeks
  The abdominal strength will be assessed by Mc Gill torso muscular endurance battery test. it consists of three endurance tests: trunk flexor, trunk lateral and trunk extensor endurance test. if holding time of these tests is more than 120 sec, core stability is interpreted as excellent.
Quality of life will be measured by SF-36 | 6 weeks
  Short-Form Health Survey (SF36) will be used to measure quality of life. It includes physical function, physical pain, general health status, energy, social function, emotional function, mental health, and indicators of health changes. scores range from 0-100. the lower the score the more disability. the higher the score the less disability.

CONTACTS AND LOCATIONS:
Overall Officials: Ujala Afzal, Principal Investigator — Foundation University Islamabad
Locations (1):
- Foundation University Islamabad, Islamabad, Federal, Pakistan